CLINICAL TRIAL: NCT00817726
Title: A Natural History Analysis of Rapid Eye Movement Sleep Behavior Disorder as Prognostic for Parkinson's Disease
Brief Title: RBD Longitudinal as Prognostic for PD
Acronym: RBD6YR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mya Schiess, Professor - Neurology, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-08-0147
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rapid Eye Movement Sleep Behavior Disorder
Keywords: Rapid Eye Movement Sleep Behavior Disorder; Parkinson's Disease; Parkinsonian Syndromes; Atypical Parkinson's; RBD; PD; fMRI; PSP; MSA
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood (serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1- RBD: polysomnographically diagnosed RBD patients. RBD is a sleep disorder diagnosed by a sleep lab in which the individual has muscle movements during the phase of deep sleep during which the muscles should be relaxed. Suspicion of RBD by history will be confirmed during screening.
- 2 - control: control:
  * must not have any neurological degenerative diagnosis.
  * must NOT have RBD.
  * must be able to age and/or gender-match to RBD and PD subjects already enrolled.

SUMMARY:
* Purpose - to validate a combination of biological and clinical markers in the rapid-eye-movement (REM) sleep behavior disorder (RBD) population as indicative of the pre-symptomatic stage of Parkinson's disease (PD).
* Procedures - All subjects (RBD diagnosis and controls) will have 1) a medical and neuro history and physical including videotape of movements, 2) neuropsychological testing, 3) a sleep study, 4) olfactory testing, 5) blood draw for serum testing , 6) functional MRI. All of these procedures are often performed clinically in the diagnosis of PD. Enrollment of subjects with PD is complete. Any testing performed prior to enrollment as part of the clinical evaluation may be used in place of repeating the procedure for the study. Subjects will be followed for 5 years. It is hypothesized that a 5 year follow up may capture a significant number of pre-Parkinson's subjects who will be diagnosed. Subjects may be offered a repeat enrollment after 5 years.

DETAILED DESCRIPTION:
Enrollment of PD and PS cohorts is complete. Currently enrolling only confirmed RBD and Controls.

ELIGIBILITY:
Inclusion Criteria:

1. 35-70 year old men & women
2. (1) Diagnosis of idiopathic RBD (see AASM criteria), 2) Normal control or control with a non-neurodegenerative disorder, age and gender-matched to (1)
3. Gives written informed consent
4. Pregnant women are not excluded, but will be identified by HCG.

Exclusion Criteria:

a A diagnosis of any non-Parkinsonian Neurodegenerative Disease.

b. Any unstable or uncontrolled medical or psychiatric condition.

c. Parasomnia or RBD not idiopathic, eg., secondary to metabolic derangement or medicine effect.

d. Renal (creatinine over 1.6) or hepatic insufficiency (LFT significantly out of range), or a history of significant uncontrolled cardiac disease.

e. Significant dementia (MMSE<25 of 30 or MOCA<25/30) that would interfere with study procedures or informed consent.

f. Any reason which, in the opinion of the PI, would increase the risk or decrease the value of any study procedure.

g. fMRI will not be performed for anyone for whom the screening questionnaire indicates is ineligible for MRI imaging.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with polysomnographically-documented RBD, non-neurodegenerative diagnosis Age and gender matched non-RBD diagnosis, non-neurodegenerative diagnosis idiopathic PD diagnosis atypical PD diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Identify the key cognitive and non-motor characteristics for early PD diagnosis | 5 years
  periodically performed set of clinical and imaging parameters suspected to be linked to PD to see if, as a group, these parameters could identify those at risk for motor symptoms of PD before these symptoms develop.

SECONDARY OUTCOMES:
Further characterize the sleep behavior patterns, olfactory function, and neurologic assessments of subjects longitudinally, over 5 years, within each group of patients. | 5 years
  perform baseline sleep study, olfactory testing and clinical neurologic exam followed by periodically performed set of clinical parameters.
functional MRI of the brain and eye tracking testing, identification of distinct features in PD | beginning of study and at 2 years
  Perform fMRI at baseline and at 2 years followed by periodically performed set of clinical parameters.
identify key fluid-based PD-associated molecular markers that identify disease state or progression | 5 years
  parameters within blood may be present & measurable well before motor symptoms of PD are seen.

CONTACTS AND LOCATIONS:
Overall Officials: Mya C Schiess, MD, Principal Investigator — The University fo texas Health Science Center at Houston
Locations (1):
- University of texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No